CLINICAL TRIAL: NCT04012983
Title: Possible Role of Gingival Crevicular Fluid Levels of Chemerin and Fibroblast Growth Factor 21 as Biomarkers of Periodontal Disease in Diabetic and Non-diabetic Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mohamed Amr, Associate Professor, Cairo University
Other Study IDs: chemerin and FGF21
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Periodontal Disease (Diagnosis); Diabetes Mellitus, Type 2
MeSH Terms: conditions — Periodontal Diseases; Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- diabetic patients with periodontitis
  Interventions: Diagnostic Test: gingival crevicular fluid level
- periodontitis patients
  Interventions: Diagnostic Test: gingival crevicular fluid level
- healthy control
  Interventions: Diagnostic Test: gingival crevicular fluid level

INTERVENTIONS:
Diagnostic Test: gingival crevicular fluid level — gingival crevicular fluid collection

SUMMARY:
The current study aims to spot the light on the possible role of gingival crevicular fluid (GCF) level of Chemerin and FGF21 to study their potential role as biomarkers of periodontal disease and to understand their role in the link between periodontitis and diabetes .

The study will be conducted on three groups; group (A) include fifteen controlled T2 DM patients suffering from periodontitis, group (B) include fifteen patients suffering from periodontitis alone, and group C) include fifteen periodontally and medically healthy individuals. GCF samples will be collected from all participants for assessment of Chemerin and FGF 21. Samples will be analysed using ELISA technique.

ELIGIBILITY:
Inclusion Criteria:

* age range between 35 and 60 years
* a minimum of 20 natural teeth.
* Type 2DM patients exhibiting HbA1c 6-8% and FPG ≥126 mg/dL for more than one year who did not complain of any systemic diseases other than t2DM
* periodontitis patients with moderate to severe periodontitis having gingival index GI ≥ 1, probing depth PD ≥ 5, and clinical attachment level CAL ≥ 4 mm, and bone loss affecting > 30% of existing teeth on clinical/radiographic examination

Exclusion criteria

* uncontrolled diabetes mellitus
* systemic diseases which may affect the biomarkers levels and the periodontal conditions.
* Exposure to steroid therapies, radiation/immune-suppressive therapies.
* Allergic reaction to any kind of drug.
* Smoking over the past 5 years.
* Periapical pathologies.
* Exposure to mechanical forces as a result of occlusion/ orthodontics.
* History of periodontal or drug therapies within the previous 6 months.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: forty five individuals (ranging in age from 35-60 years) recruited from the outpatient clinic of Oral Medicine, and Periodontology Department, Faculty of Dentistry, Cairo University
  The participants were divided into the following three groups:
  Group (1): 15 patients with periodontitis and controlled t2DM and no other systemic disease.
  Group (2): 15 systemically healthy individuals having periodontitis. Group (3): 15 periodontally and systemically healthy individuals.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
measurement of the level of FGF21 (pg/ml) in gingival crevicular fluid of diabetic patients with periodontitis | baseline
  assessment of GCF FGF21 in diabetic patients with periodontitis
measurement of the level of FGF21 (pg/ml) in gingival crevicular fluid of periodontitis patients | baseline
  assessment of GCF FGF21 in patients with periodontitis
measurement of the level of FGF21 (pg/ml) in gingival crevicular fluid of healthy controls | baseline
  assessment of GCF FGF21 in healthy individuals

SECONDARY OUTCOMES:
measurement of the level of chemerin (ng/ml) in gingival crevicular fluid of diabetic patients with periodontitis | baseline
  assessment of GCF chemerin in diabetic patients with periodontitis
measurement of the level of chemerin (ng/ml) in gingival crevicular fluid of periodontitis patients | baseline
  assessment of GCF chemerin in patients with periodontitis
measurement of the level of chemerin (ng/ml) in gingival crevicular fluid of healthy controls | baseline
  assessment of GCF chemerin in healthy individuals

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided